CLINICAL TRIAL: NCT05916235
Title: Photobiomodulation for Management of Temporomandibular Disorder Pain
Acronym: ULLTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202300986; UG3DE030433-01A1 (NIH); UH3DE030433 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pain Related to TMD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: Active PBM (Experimental): PBM has been used clinically in the treatment of musculoskeletal and other pain conditions for over 30 years. Despite the low quality of the existing evidence, PBM has been increasingly used in other countries for the treatment of TMD. However, in the US PBM is not widely used for the treatment of TMD pain. Due to the multifactorial nature of chronic TMD pain, we propose that a multimodal PBM protocol targeting multiple pathophysiological mechanisms will be the optimal approach for PBM implementation in patients with TMD.
  Interventions: Device: THOR® laser system
- Sham PBM (Sham Comparator): When applying PBM therapy, there are some heating elements in the treatment device, and most of the sham treatment devices available do not offer this feature, which increases the likelihood of unblinding both the patient and the interventionist. The THOR® LX2.3 PBM machine includes this new feature, such that the sham condition mimics the heating activity of the active treatment.
  Interventions: Device: THOR® laser system

INTERVENTIONS:
Device: THOR® laser system — We chose the THOR® laser system given because their active treatment arm uses both coherent laser and monochromatic LED light. Therefore, we will use three types of active probes in this investigation including, A) Single Laser 810 NM 200 mw; B) Laser Cluster of 810 NM equivalent to 1 WATT and; C) LED Cluster, 34 X 660nm at 10 mw and 35 850nm, 30mw 1390mw total. As detailed in Table 3. We propose to use these three PBM probes in concert for the treatment of TMD pain. Laser A (Single Diode Laser) is designed for isolated trigger points and superficial muscles. Laser B (Cluster Laser) is designed for a more diffuse treatment area,targeting analgesia, anti-inflammatory, and deep tissue repair. Laser C (LED Cluster) is purportedly designed for the presence of diffuse inflammation.

SUMMARY:
Photobiomodulation (PBM), is FDA-approved for temporary relief of muscle and joint pain, but there is no indication for TMD. Our goal in this study is to conduct a clinical trial of multimodal PBM for TMD pain. This study will be a double-blind, sham-controlled, randomized trial testing the efficacy of PBM for pain related to TMD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and older
* Meets the CATI pre-screening criteria during pre-screening visit [participant-reported facial pain for at least 3 months and an average pain intensity rating for the week preceding CATI of ≥30 on a numerical rating scale (NRS, 0-100)].
* Willing to provide signed and dated informed consent
* Willing to to comply with all study procedures and to be available for the duration of the study
* Meets diagnostic criteria for TMD (Masticatory Muscle disorder, 1 A: Myalgia) during Visit 0
* Completes a minimum of 4 of 7 daily symptom diary (DSD) entries prior to Visit 1 (Randomization visit), and the weekly average pain score on this DSD is ≥30 of 100

Exclusion Criteria:

* Active rheumatologic disease
* Has a medical condition, laboratory finding, or physical exam finding (e.g., renal failure or dialysis, uncontrolled diabetes mellitus, or uncontrolled seizures) that precludes participation as determined by the investigator
* Initiated occlusal appliance therapy within 30 days prior to CATI
* Initiated non-pharmacologic therapy, such as acupuncture, biofeedback, and/or TENS within 30 days prior to CATI
* Is in active orthodontic treatment
* Received any injection therapy (e.g., tender or trigger point injections, steroid injections) for the management of pain within 14 days prior to the CATI
* Has a history of facial trauma or orofacial surgery within 6 weeks prior to CATI
* Has a history of psychiatric hospitalization within one year prior to CATI
* Currently pregnant or lactating
* Has a known hypersensitivity to laser therapy
* Currently being treated with chemotherapy or radiation therapy
* Is undergoing treatment with another investigational drug or treatment initiated within 30 days prior to the Screening and Baseline Visit
* Initiated a new daily prescribed or over-the counter medication for the management of pain within 30 days prior to Screening and Baseline Visit.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study as determined by the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Pain Level Change with PBM treatment using a Numerical Rating Scale | Through study completion; about 6 months
  The primary outcome measure will be the average of daily pain ratings on the numerical rating scale (0 = no pain, 100 = worst pain imaginable) from the Daily Symptom Diary. Daily pain ratings averaged over one week prior to randomization will be treated as the baseline variable. The average daily pain for one week prior to Visit 9 will be treated as the primary endpoint. This outcome measure averaged across multiple days provides a stable measure of pain that is less subject to recall bias.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rodriguez MG, Warchol M, Rubio S, Cabrera P, Reever R, Hosney S, Migliorati CA, Gibson Iii FC, Ohrbach R, Fillingim RB, Wallet S, Ribeiro Dasilva MC. In vitro effects of dual wavelength photobiomodulation on monocytic response in painful temporomandibular disorder. J Oral Facial Pain Headache. 2025 Dec;39(4):252-257. doi: 10.22514/jofph.2025.082. Epub 2025 Dec 12. PMID 41436122
- [Derived] Rubio S, Cabrera P, Reever R, Migliorati C, Ohrbach R, Gibson FC 3rd, Li Z, Mickle A, Conic RRZ, Fillingim RB, Ribeiro Dasilva M. A protocol for a randomized controlled trial of photobiomodulation for management of temporomandibular disorder pain in Adults. Contemp Clin Trials Commun. 2025 Nov 24;48:101571. doi: 10.1016/j.conctc.2025.101571. eCollection 2025 Dec. PMID 41399628